CLINICAL TRIAL: NCT04153695
Title: Therapeutic Flamenco Musical Intervention in Pregnant Women
Brief Title: Flamenco Music Therapy in Pregnant
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Telethusa Centre for Flamenco Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TelethusaFlamenco
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Pregnancy; Music; Therapy
Keywords: Pregnant; Anxiety; Depression.; Flamenco music
MeSH Terms: conditions — Anxiety Disorders; Depression | interventions — Music Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): To listen flamenco music during 30 minuts per day, during 2 weks
  Interventions: Other: Music Therapy
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Music Therapy — to listen flamenco music during 30 minuts per day during 2 weeks
  Arms: Experimental

SUMMARY:
The use of music as a therapy for the psychological and emotional improvement of pregnant women has been well studied. Our hypothesis is that flamenco music can also involve psycho-emotional improvements in pregnant women

DETAILED DESCRIPTION:
The objective of the study is to analyze the effects of a flamenco musical intervention on the stress and anxiety of pregnant women in five Management Units of the Sanitary District in Bahía de Cádiz-La Janda (Spain).

50 pregnant women will voluntarily participate in this study (25 in a control group and 25 in the experimental group) The psychological health assessment will be measured through the Perceived Stress Scale (PSS), the State-Trait Anxiety Inventory (S-STAI) and the Edinburgh Postnatal Depression Scale (EDPS) pre and post exposure.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer
* Single pregnancy
* Uncomplicated pregnancy,
* Expectations of vaginal delivery without complications
* Gestational age between 18 and 33 weeks,

Exclusion Criteria:

* Visual disorders
* Hearing disorcers
* Mental or cognitive disorders
* Difficulties in pregnancy,
* Medical complications,
* Smoker during the gestation period

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2019-12-19 (Estimated); Study Completion 2020-01-25 (Estimated)

PRIMARY OUTCOMES:
Perceived Stress Scale | 4 months
  Perceived Stress Scale is used in order to measure anxiety in adults. It clearly differentiates between the temporary condition of "state anxiety" and the more general and long-standing quality of "trait anxiety". It consists of fourteen questions that refer to the feelings and thoughts of the person surveyed during the last month.
  It consists of fourteen questions that refer to the feelings and thoughts of the person surveyed during the last month. The answer format of each question is a Likert scale with five possible options. The minimum value is 0 (never) and maximun is 4 (very often). Higher score means the worse outcome.
State-Trait Anxiety Inventory | 4 months
  It is a psychological inventory based on a 4-point Likert scale (from 0 or "Almost Never" to 3 or "Almost Always") and it consists of 20 questions on a self-report basis. The STAI measures two types of anxiety - state anxiety, or anxiety about an event, and trait anxiety, or anxiety level as a personal characteristic. Higher scores are positively correlated with higher levels of anxiety, so the worse outcome.
Edinburgh Postnatal Depression Scale | 4 Months
  The Edinburgh Postnatal Depression Scale is a set of 10 screening questions that can indicate whether a parent has symptoms that are common in women with depression and anxiety during pregnancy and in the year following the birth of a child. This is not intended to provide a diagnosis - only trained health professionals should do this.
  Each question has four items and is evaluated from 0 to 3, according to the increase in the severity of the symptom. Questions 3, 5, 6, 7, 8, 9, 10 rank in reverse order. The total score can range from 0 to 30, with 0 being the best result and 30 the worst.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Vargas-Macías, PhD, Principal Investigator — Telesthusa Centre for Flamenco Research
Locations (1):
- Alfonso Vargas-Macías, Cadiz, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Website of the Research Project — http://www.flamencoinvestigacion.es/pi-a5-2019-musica-flamenca-embarazadas/